CLINICAL TRIAL: NCT03004118
Title: Therapeutic Effect of Ursodeoxycholic Acid on Duodenal Permeability and Meal Related Sensory Motor Function in Functional Dyspepsia Patients
Brief Title: Therapeutic Effect of Ursodeoxycholic Acid in Functional Dyspepsia
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UDC1
Record Dates: First submitted 2016-12-05; First posted 2016-12-28 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Ursodeoxycholic Acid; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ursochol (Active Comparator): About 10.5mg/kg/day of ursochol (calculated before start study for each participant individually) (combination of ursochol 150 and 300) divided in 2 doses per day (during lunch and dinner). Oral intake. Tablets. 4 weeks.
  Interventions: Dietary Supplement: Nutridrink; Device: High resolution manometry probe; Device: perfusion catheter; Drug: Ursochol oral tablet; Device: Duodenal fluid aspiration catheter; Procedure: Duodenogastroscopy; Procedure: Blood sample
- Placebo (Placebo Comparator): Same amount of pills as ursochol (calculated before start study for each participant individually) divided in 2 doses per day (during lunch and dinner). Oral intake. Tablets. 4 weeks.
  Interventions: Dietary Supplement: Nutridrink; Device: High resolution manometry probe; Device: perfusion catheter; Drug: Placebo Oral Tablet; Device: Duodenal fluid aspiration catheter; Procedure: Duodenogastroscopy; Procedure: Blood sample

INTERVENTIONS:
Dietary Supplement: Nutridrink — Liquid meal of 200ml
Device: High resolution manometry probe — Catheter inserted via the nose into the stomach to measure intragastric pressure.
Device: perfusion catheter — Catheter inserted via the nose into the stomach to perfuse the nutridrink intragastricly.
Drug: Placebo Oral Tablet — 4 week oral intake (daily)
  Arms: Placebo
Drug: Ursochol oral tablet — 4 week oral intake (daily) (dose of 10.5mg/kg/day)
  Arms: Ursochol
Device: Duodenal fluid aspiration catheter — Catheter inserted via the nose into the duodenum to aspirate duodenal fluids for 2.5 hours.
Procedure: Duodenogastroscopy — Catheter inserted via the mounth into the duodenum to take duodenal biopsies.
Procedure: Blood sample — Blood sample will be taken to measure liver enzyme serum levels and marker for bile acid synthesis.

SUMMARY:
The investigators aim to evaluate ursochol as a therapy in functional dyspepsia. The objectives of the study are to evaluate the effect of ursochol on duodenal permeability and dyspeptic symptoms and on duodenal low-grade inflammation, bile acid composition, bile acid receptor expression, nutrient tolerance and intragastric pressure.

Cross-over, controlled, randomized, double blinded, placebo-controlled trial with a 4 week intake of ursodeoxycholic acid (ursochol) versus a 4 week intake of placebo and a 4 week washout period in between. Two study days are planned during week 4 and week 12. During the 14 weeks, the patients have to fill in a diary. And for 14 weeks in total, the patients have to discontinue intake of proton pump inhibitors, drugs effecting gastric motility and NSAIDs and replace their oral anticonception with non-oral anticonception. Every two weeks of the study the investigator will call the participants to see how they are/if they have any discomforts or side effects.

DETAILED DESCRIPTION:
Functional dyspepsia patients will be recruited and screened for inclusion in the study. The participants will be asked to not take proton pump inhibitors, drugs effecting gastric motility and NSAIDs and oral anticonception for fourteen weeks. First, they will stop with their daily drug intake of PPIs and NSAIDs for two weeks, then they will take placebo or UDC for four weeks, two doses every day during lunch and dinner. Afterwards, there will be a washout period of four weeks, and again four weeks of UDC or placebo intake. The patients will receive a diary in which they describe their symptoms/discomforts every day for 14 weeks. All participants and the investigator will be blinded to the nature (UDC or placebo) of the pills. The random order in which a certain patient gets his pills has been decided by the pharmacy of UZ Leuven and is also unknown for the investigator (double blinded). During week two, four, six, eight, ten and twelve we will have a phone conversation with the patients to discuss their symptoms/discomforts.

During week four and week twelve, the patients will come to the hospital for one day after an overnight fast. First, they are asked to fill in a bundle of questionnaires concerning physical complaints, depression, anxiety (disturbances), pain/disease, body/interoceptive awareness, trauma/abuse and personality and to give a fecal sample that they've collected the day before. The fecal sample will be used to evaluate the gastrointestinal microbiota in FD patients. Then, two blood samples, to evaluate liver function parameters and bile acid synthesis, will be taken and an endoscopy will be performed. All endoscopies will be performed by an experienced endoscopist (Jan Tack) and nine duodenal biopsies (2 biopsies at a time) (Radial Jaw™3 with needle; outside diameter 2.2mm; Boston Scientific, 302 Parkway, Global Park, Heredia, Costa Rica) will be obtained. To measure the in vitro transepithelial resistance, 3 biopsies will be examined using an adapted mini-Ussing chambers system. After equilibration, the mucosal side of the tissue will be exposed to 4kDa FITC-dextran as a measure of paracellular permeability. A sample will be taken from the serosal side during 2h at 30min interval. The concentration of fluoresceïn will then be measured using a fluorescence plate reader. Also, two biopsies will be used for mRNA extraction and subsequent cDNA synthesis. This cDNA will be used to measure the gene expression of bile acid receptors by means of real-time RT-PCR. In addition, one biopsy will be prepared for immunohistochemistry and two will be used for western blot to measure changes in distribution/expression of the bile acid receptor proteins. One biopsy will be obtained to study ultrastructural alterations by transmission electron microscopy.

After the endoscopy, an aspiration catheter will be positioned in the duodenum. The position of the catheter will be briefly checked by fluoroscopy (typically 2-3 seconds, however never more than 15 seconds). After positioning of the catheter, it is fixed to the subject's chin and he/she is asked to take place in a chair for the remainder of the experiment. For one hour, every 15 minutes duodenal fluids will be collected during fasted state. Next, a high resolution manometry catheter (HRM) will be placed in the gastric fundus to measure intragastric pressure and a perfusion tube (OD 2 mm) will be introduced through the nose and positioned in the stomach. After positioning of the catheters, they are fixed to the subject's chin and he/she is asked to take place in a chair for the remainder of the experiment. After a stabilization period of 15 minutes, intragastric infusion of the nutrient drink (Nutridrink, Nutricia; 630 KJ, 6 g proteins, 18.4 g carbohydrates, and 5.8 g lipids per 100 mL) will start at a constant speed of 60 mL per minute (determined by an automated system using a peristaltic pump). Intragastric pressure will be measured with a 36-channel high resolution manometry system, through the intragastric manometry probe. At 1-minute intervals, the subjects will be asked to score their satiation using a graphic rating scale that combines verbal descriptors on a scale graded 0-5. At 5-minute intervals the volunteers will be asked to fill out a VAS for 11 dyspeptic symptoms. The intragastric infusion will be stopped as soon as the volunteers score maximally on one of the 11 epigastric symptoms or when a score of 5 is reached on their satiety scores. 10 minutes thereafter, the catheters will be disconnected and removed. After the nutrient drink infusion, duodenal fluids will be collected every 15 minutes for 1.5 hour during fed state. Finally, the last catheter is removed and the volunteer can go home.

ELIGIBILITY:
Inclusion Criteria:

Men and women (age 18-60 years) who meet the Rome IV criteria for functional dyspepsia can participate in the study. For 14 weeks, patients need to discontinue their intake of proton pump inhibitors, drugs effecting gastric motility and NSAIDs. If a female participant takes oral anticonception, she has to switch to non-oral anticonception for this study. All participants will receive and sign a copy of the informed consent.

Exclusion Criteria:

* refused informed consent
* pregnant women or women who are breastfeeding
* diabetes mellitus
* celiac disease
* coagulation disorders/anticoagulant therapy
* not well functioning liver and gallbladder
* active stomach or gut ulcer
* biliary colic, calcified gallstones
* acute infection of gallbladder or bile ducts, bile duct obstruction
* intestinal disorders such as ulcerative colitis, Crohn's disease
* lactose intolerance
* allergies/sensitivity (asthma, allergic to bile acids, eczema, allergic rhinoconjunctivitis)
* Intake of oral anticonception, barbiturates, antacid, colestyramine or colestipol, nitrendipine, cyclosporine, ciprofloxacine, rosuvastatine.
* first degree relatives with celiac disease, Crohn's disease or type I diabetes mellitus Severe kidney malfunction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Duodenal mucosal transepithelial electrical resistance (TEER) (Ohm*cm^2) measured with adapted ussing chamber system | 2 hours
  Transepithelial resistance is a measure for mucosal integrity
Duodenal mucosal paracellular passage of Fitc Dextran 4kDa (pmol) measured with FLUOstar Omega microplate reader. | 2 hours
  Paracellular permeability is a measure for mucosal integrity
Dyspeptic symptom occurence and intensity during meal intake via questionnaire every 1 minute until end of the meal | About 10 minutes
  Scoring of dyspeptic symptom occurence by patients during nutrientdrink perfusion
Daily occurence and intensity of dyspeptic symptoms via LPDS diary | 14 weeks
  Leuven Postprandial Distress Scale, a questionnaire for symptom assessment in the functional dyspepsia/postprandial distress syndrome.

SECONDARY OUTCOMES:
Glycocholic acid concentration (mM) | 14 weeks
  Bile salt
Taurocholic acid concentration (mM) | 14 weeks
  Bile salt
Glycochenodeoxycholic acid concentration (mM) | 14 weeks
  Bile salt
Taurochenodeoxycholic acid concentration (mM) | 14 weeks
  Bile salt
Glycodeoxycholic acid concentration (mM) | 14 weeks
  Bile salt
Taurodeoxycholic acid concentration (mM) | 14 weeks
  Bile salt
Glycoursodeoxycholic acid concentration (mM) | 14 weeks
  Bile salt
Tauroursodeoxycholic acid concentration (mM) | 14 weeks
  Bile salt
Protein expression of duodenal bile acid receptor VDR | 14 weeks
  Western blot
Protein expression of duodenal bile acid receptor FXR | 14 weeks
  Western blot
Protein expression of duodenal bile acid receptor PXR | 14 weeks
  Western blot
Protein expression of duodenal bile acid receptor TGR5 | 14 weeks
  Western blot
Protein expression of duodenal bile acid receptor CAR | 14 weeks
  Western blot
RNA expression of duodenal bile acid receptor VDR | 14 weeks
  Real time RT-PCR
RNA expression of duodenal bile acid receptor FXR | 14 weeks
  Real time RT-PCR
RNA expression of duodenal bile acid receptor PXR | 14 weeks
  Real time RT-PCR
RNA expression of duodenal bile acid receptor TGR5 | 14 weeks
  Real time RT-PCR
RNA expression of duodenal bile acid receptor CAR | 14 weeks
  Real time RT-PCR
Intragastric pressure measurement via an high resolution manometry (HRM) probe | 1 hour
Mast cell count in duodenal biopsies (number of mastcells/ mm^2 lamina propria) | 14 weeks
Eosinophil count in duodenal biopsies (number of eosinophils/ mm^2 lamina propria) | 14 weeks

IPD SHARING:
Plan to Share IPD: No